CLINICAL TRIAL: NCT06704867
Title: High Flow Nasal Cannula Compared to Standard Oxygen Therapy for Endoscopic Ultrasound Procedure in High Risk Patients on Recovery Time and Procedural Conditions
Brief Title: High Flow Nasal Cannula Compared to Standard Oxygen for Endoscopic Ultrasound
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Principal Investigator, Bhargavi Gali, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24-003924
Record Dates: First submitted 2024-11-20; First posted 2024-11-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Endoscopic Ultrasound
Keywords: High Flow Nasal Cannula; High BMI; Oxygen

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard oxygen therapy (No Intervention): Standard oxygen therapy will be initiated utilizing 2-4 liters of oxygen with a nasal cannula.
- High Flow Nasal Cannula (Experimental): A high flow oxygen device with 100% FiO2 will be initiated prior to endoscopic ultrasound.
  Interventions: Other: High flow nasal cannula

INTERVENTIONS:
Other: High flow nasal cannula — Subjects undergoing endoscopic ultrasound will receive high flow nasal cannula during the procedure
  Arms: High Flow Nasal Cannula

SUMMARY:
The purpose of the study is to evaluate the use of high flow nasal cannula versus standard oxygen therapy for high-risk patients undergoing endoscopy procedures.

DETAILED DESCRIPTION:
Patients with a higher BMI are at greater risk for lower oxygen levels which can delay the endoscopy procedure. This research is being conducted to find out if high risk patients will have a shorter recovery time and improved procedural conditions with a high flow nasal cannula versus standard oxygen therapy.

ELIGIBILITY:
Inclusion Criteria:

• All patients age 18 years and older who present to Gonda 2 procedural area for Endoscopic ultrasound (EUS) with or without endoscopy (EGD)/biopsy/tissue sampling. with BMI ≥ 35 kg/m2 (BMI within the past 6 months in electronic medical records or at current procedure) who are able to consent will be approached for potential enrollment.

Exclusion Criteria:

* Need for general anesthesia for the procedure instead of the standard monitored anesthesia care.
* Patients undergoing combined procedure: Therapeutic EUS/combined procedures including EUS/ERCP, EUS/colonoscopy
* Patients on home oxygen therapy, or the diagnosis of "severe COPD"
* Patients with existing tracheostomy
* Inpatients undergoing EUS
* Inability to consent
* Cognitive impairment
* Blocked nasal passages
* Trauma/previous surgery to the nasopharynx
* Irregularities of the nose, face, or airway such that HFNC cannot be properly fitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Decrease recovery time | 4 hours
  Time measured in minutes for participants to enter post anesthesia care until the nurse marks "ready for discharge" in the medical record.

SECONDARY OUTCOMES:
Improve procedural conditions | 1 hour
  Decreased number of times the procedure is paused or delayed.

CONTACTS AND LOCATIONS:
Overall Officials: Bhargavi Gali, MD, MHA, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No